CLINICAL TRIAL: NCT01948752
Title: Clinical Trial of Menu Labeling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Waterloo (Other)
Collaborators: Canadian Cancer Society (CCS) (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Uwaterloo
Record Dates: First submitted 2013-04-17; First posted 2013-09-24 (Estimated); Last update posted 2013-09-24 (Estimated); Status verified 2013-09

CONDITIONS: Calorie Consumption
Keywords: Nutrition policy; food labelling; diet; obesity; health behavior
MeSH Terms: conditions — Obesity; Health Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Menu - no nutrition information (control) (No Intervention): Participants were randomized to receive one of four menus that each contained different type of nutrition information. This condition included a "normal" menu with no nutrition information.
- Calorie labels (Experimental): Participants were randomized to receive one of four menus that each contained different type of nutrition information. This condition included menus with the calorie amounts displayed.
  Interventions: Other: Nutrition information on menus
- Calorie Traffic Light (Experimental): Participants were randomized to receive one of four menus that each contained different type of nutrition information. This condition included menus with calorie amounts in green/amber/red "traffic lights" to signify low/medium/high amounts.
  Interventions: Other: Nutrition information on menus
- Multi-Traffic Light (Experimental): Participants were randomized to receive one of four menus that each contained different type of nutrition information. This condition included menus with calorie amounts as well as sodium, fat, and sugar amounts in green/amber/red "traffic lights" to signify low/medium/high amounts.
  Interventions: Other: Nutrition information on menus

INTERVENTIONS:
Other: Nutrition information on menus
  Arms: Calorie Traffic Light; Calorie labels; Multi-Traffic Light

SUMMARY:
The current study sought to examine the effect of menu labeling on food ordering and food consumption, including the effect of displaying calories along with other nutrients, such as sodium, fat, and sugar, as well as in different formats, such as traffic lights.

The investigators hypothesize significant differences in the calorie amount of menu selections and food consumption across experimental conditions. The investigators anticipate that calorie amounts will be significantly higher in the no calorie information) compared to each of the other 3 conditions, and significantly lower in the Traffic Light conditions compared to calories only condition.

2) Individuals in Condition 1 (no calorie information) will be significantly more likely to underestimate the calorie content of their meals compared to individuals in the intervention conditions.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older,
* able to speak and read English

Exclusion Criteria:

- no food allergies to gluten or other grain products

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 661 (Actual)
Dates: Start 2010-11; Primary Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Calorie consumption. | Calorie consumption was recorded for the meal consumed during the visit to the laboratory, approximately 30 minutes after the start of the study. No additional follow-up was conducted after the laboratory visit.
  Participants consumed the food during the study visit, after ordering from the menus and completing survey measures. The calorie content of all food and beverage items ordered by each participant was calculated immediate after the study session using information provided by Subway. All items were weighed immediately prior to delivery to participants. After participants indicated that their meal was completed, research assistants collected and weighed any leftover food or beverage portions. A consumption variable was calculated for calorie, fat, sodium, and sugar consumption for each participant by subtracting the estimated number of calories in food and beverage waste from the total for the meal, based on differences in weight. No measures were collected after the study visit.

SECONDARY OUTCOMES:
Calorie content of meals ordered by participants. | Calorie content was recorded for the meal consumed during the visit to the laboratory, approximately 30 minutes after the start of the study. No additional follow-up was conducted after the laboratory visit.
  Calorie content of the meal consumed during the laboratory visit was subsequently calculated using nutrition data for each food and beverage item.

CONTACTS AND LOCATIONS:
Overall Officials: David Hammond, PhD, Principal Investigator — University of Waterloo
Locations (1):
- School of Public Health, University of Waterloo, Waterloo, Ontario, Canada

REFERENCES:
- [Derived] Hammond D, Goodman S, Hanning R, Daniel S. A randomized trial of calorie labeling on menus. Prev Med. 2013 Dec;57(6):860-6. doi: 10.1016/j.ypmed.2013.09.020. Epub 2013 Oct 7. PMID 24113263